CLINICAL TRIAL: NCT07273149
Title: A Decentralised, Open-labelled, Clinical Study to Assess the Effectiveness of a Marketed Denture Adhesive in Food Occlusion in Denture Wearers in a Real-world Setting
Brief Title: A Study to Assess the Effectiveness of a Marketed Denture Adhesive in Real-World Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 400027
Record Dates: First submitted 2025-11-28; First posted 2025-12-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Denture Retention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- No Adhesive Use Followed by Adhesive Use (Experimental): Participants will wear their dentures without any denture adhesive cream for 3 weeks from Day 1 to Day 21 of the study. Participants will wear their dentures with the denture adhesive cream (Poligrip Power Max Hold + Seal) as per the label instructions, once daily for 3 weeks from Day 22 to Day 42 of the study.
  Interventions: Device: Poligrip Power Max Hold + Seal

INTERVENTIONS:
Device: Poligrip Power Max Hold + Seal — Poligrip Power Max Hold + Seal denture adhesive cream containing sodium-calcium mixed partial salt of poly(methylvinylether/maleic acid) and carboxymethylcellulose.

SUMMARY:
The purpose of this decentralised study in a real-world setting is to assess the effectiveness of a marketed denture adhesive (Poligrip Power Max Hold + Seal) in preventing food entrapment under dentures (self-assessed). The study will evaluate participants perceived food occlusion of a marketed denture adhesive over three weeks compared to no adhesive use over three weeks in a real-world setting.

DETAILED DESCRIPTION:
This will be an open-labelled, decentralised, 6-week study to assess the effectiveness of food occlusion of a marketed denture adhesive in healthy partial and/or full denture wearers aged 18 and above in a real-world setting. Study comprises of 3 weeks of no adhesive use (Day 1 to 21) followed by 3 weeks of adhesive use (Day 22 to 42). Participants will complete Daily Food Occlusion Questions for 3 weeks without using adhesive cream and another 3 weeks with using adhesive cream. Sufficient participants will be screened to enroll approximately 375 participants to ensure that around 300 of these participants will successfully complete the entire study. Participants will be recruited through digital platforms through pre-screening questionnaires followed by a screening virtual visit.

ELIGIBILITY:
Inclusion Criteria:

* Participant's provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participants from all genders (male, female, not specified).
* Participant who, at the time of screening is 18 years old and above.
* Participants who are willing and able to comply with all study related activities as shown in the schedule of activities, study restrictions, and other study procedures.
* A participant in good general and mental health with no self-reported clinically significant or relevant abnormalities in medical history or upon a previous oral examination, or condition, that would impact on the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* A participant who is a habitual wearer of partial or full denture defined as participant who wear their dentures for the majority of their time whilst awake.
* Participants should have a relatively well-fitted denture (self-assessed).
* Participants who reside in the United States (except for Hawaii and Alaska).

Exclusion Criteria:

* An employee either directly involved in the conduct of the study or a member of their immediate family; or an employee of Lindus Health otherwise supervised by the investigator; or, a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant who has been previously enrolled in this study.
* Participants who have a clinical condition as self-reported on the screening questionnaire, which include:

  1. Participants who have undergone treatment for periodontal or gum disease within 6 months of screening or are currently undergoing treatment for periodontal or gum disease.
  2. Participants who have been informed by Health Care Professional (HCP) that they have active periodontitis.
  3. Participants who have been informed by HCP that they have active candida infection.
  4. Participants who have been informed by HCP that they have active caries.
  5. Participants with any chronic and/or severe painful health condition(s) which lead to regular use of pain relief medications more than 3 days a week.
  6. Participants who have any clinically significant or relevant oral abnormality (example, temporomandibular joint problems) or palate problem that could have impact on their participation in the study.
  7. In the opinion of the investigator, participants with an acute or chronic medical or psychiatric condition or laboratory abnormality that may impact their safety, ability to follow study procedures or integrity of the study.
* A participant who is diagnosed with xerostomia or is taking any medication that is causing xerostomia.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant who has a recent history (within the last year) of alcohol or other substance abuse.
* A participant who has history of swallowing difficulties or choking.
* Participants must not receive any denture-related adjustments or treatments that alter fit, comfort or structure of their denture during the study.
* Currently taking or have taken a bisphosphonate drug (that is., Fosamax, Actenol, Boniva).
* A participant who reports a planned surgery during the study duration.
* A participant who, in the opinion of the investigator or delegate, should not participate in the study.
* A participant who is unable to read and understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Mean Score of the Food Occlusion Question Assessed Using the Numerical Rating Scale (NRS) | Up to Week 6
  Participants will answer specific food related question on a daily basis throughout the study. Participants scored the Food Occlusion Question using the NRS.

SECONDARY OUTCOMES:
Mean Daily Responses of Full-day Food Occlusion Question | Up to Week 6
  Participants will answer the Food Occlusion Question related to occlusion of food particles under denture using a Yes/No response.
Mean Food Particle Bothersomeness Score of Food Occlusion Question Assessed Using the NRS | Up to Week 6
  Participants will answer specific food related question on a daily basis throughout the study using the NRS.
Mean Comfort Score of Food Occlusion Question Assessed Using the NRS | Up to Week 6
  Participants will answer specific food related question on a daily basis throughout the study using the NRS.

CONTACTS AND LOCATIONS:
Locations (1):
- Lindus Health (virtual site), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary and key secondary endpoints and the safety data for the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.